CLINICAL TRIAL: NCT03330249
Title: Phase II Randomized Trial Comparating Two Concomitant Administration of Radiotherapy With Cisplatin in Patients With Not Operated or Inoperable HNSCC or With Recurrence High Risk in Adjuvant Postoperative Treatment
Brief Title: Comparison of Two Concomitant Administration of RT With Cisplatin in Standard Infusion or Fractional Infusion
Acronym: CisFRad
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC 2015-02
Record Dates: First submitted 2017-01-17; First posted 2017-11-06 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Split Cisplatin and radiotherapy (Experimental): 25 mg/m2/day IV infusion at D1 to D4, at D22 to D25, at D43 to D46 during the radiotherapy
  Interventions: Drug: Split Cisplatin; Radiation: Radiotherapy
- Cisplatin and radiotherapy (Active Comparator): 100 mg/m2/day IV infusion at D1, D22 and D43 during the radiotherapy
  Interventions: Drug: Cisplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Split Cisplatin — 25 mg/m2/day IV infusion at D1 to D4, at D22 to D25, at D43 to D46 during the radiotherapy.
  Other Names: Cisplatin infusion
  Arms: Split Cisplatin and radiotherapy
Drug: Cisplatin — 100 mg/m2/day IV infusion at D1, D22 and D43 during the radiotherapy.
  Other Names: Cisplatin infusion
  Arms: Cisplatin and radiotherapy
Radiation: Radiotherapy — 70 Gy in 35 fractions of 2 Gy in non-operated patients and 66 Gy in 33 fractions in post-operative.
  Other Names: Radiotherapy IMRT with possibly integrated boost

SUMMARY:
The general aim is to compare the cumulative dose of cisplatin administered concomitantly with radiotherapy in reference arm A (cisplatin 100 mg / m2 day 1 every 21 days) and in the experimental arm B (Cisplatin split 25 mg / m2 / J D1 to D4 all 21 days).

DETAILED DESCRIPTION:
The standard treatment for squamous cell carcinoma of the head and neck locally advanced non-operated or non-operable is a combination of radiotherapy and concomitant chemotherapy. Indeed, the meta-analysis MACH showed for RT / CT associations an absolute survival benefit of 8% compared with radiotherapy alone. Cisplatin delivered optimally, ie at a dose of 100 mg / m2 on day 1, D22 and D43 of radiotherapy is as effective as combinations of cisplatin and 5-fluorouracil.

In post operative, treatment of high risk recurrence forms by Cisplatin, concomitantly with radiotherapy, also increases local control and overall survival.

However, it is an association whose toxicity is significant. The usual limiting toxicities were mucositis, dysphagia, nausea and vomiting with malnutrition and biologically kidney failure and myelotoxicity. Only 2/3 of the patients receive 3 cycles of cisplatin initially programmed.

As shown in the RTOG 0129 trial, the number of cycles of cisplatin and thus the cumulative dose of cisplatin administered concurrently with radiation therapy, significantly influences the locoregional control, progression free survival and overall survival.

One method of reducing the toxicity and thereby, increase the cumulative dose, would be to split the administration of cisplatin.

Moreover, the efficacy of Cisplatin, which only the free fraction is active, seems correlated with AUC that peak plasma which would in turn responsible for toxicity. The completion of a pharmacokinetic study comparing the AUC and Cmax obtained with cisplatin 100 mg / m2 and cisplatin fractionated is essential.

Finally, the limiting renal toxicity induced by cisplatin is currently diagnosed using the creatinine clearance. The Neutrophil gelatinase-associated lipocalin (NGAL) urinary is a new diagnosis and prognosis marker of renal impairment following treatment with cisplatin. However, further studies are needed to validate its clinical utility.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell carcinoma of head and neck cancer stage III or IV: oral cavity, oropharynx, larynx or hypopharynx.
* Patient non-operated and / or inoperable for reasons of non extirpabilité, local and regional expansion, general state or medical condition Or
* Patient operated within 8 weeks before radiation therapy with a high risk of recurrence: unsatisfactory surgical margins (R1) and / or lymph node involvement with capsular rupture.
* Activity Index according to WHO ≤ 2
* Age ≤ 70 years
* Ventricular ejection fraction left retained> 50%
* Renal allowing the administration of cisplatin: creatinine clearance> 60 ml / min (Cockroft formula)
* Hematologic function allowing administration of CT: PNN> 1500, Pl> 100000, Hb> 9g
* Satisfactory Liver function: SGOT and SGPT <3N; total bilirubin <20 mg / dL; INR <1.5; albumin> 30 g / l
* Stomatological care adapted
* Signature of informed consent
* Bilateral neck irradiation Indication
* Women and men of reproductive age should have accepted a medically effective contraception during the treatment period and at least 6 months after discontinuation of study treatment. If pregnancy is declared by a patient or partner of a patient, it must be followed for know the evolution of pregnancy.

Exclusion Criteria:

* Cancers of the nasopharynx, sinus or nasal cavities
* Histology other than squamous
* Presence of distant metastases
* Prior systemic chemotherapy (neoadjuvant)
* Other concomitant cancer therapies
* Presence of infection requiring the use of IV antibiotics including tuberculosis and HIV infection
* Coronary insufficiency, cardiac arrhythmias, uncontrolled or symptomatic heart failure
* Uncontrolled hypertension
* Peripheral neuropathy grade> 1
* Vaccination against yellow fever and phenytoin recent or planned
* History of cancer within 5 years prior to trial entry other than cutaneous basal cell carcinoma in situ or cervical
* Pregnant woman capable of being or during lactation
* Persons deprived of liberty, under guardianship
* Inability to submit to medical monitoring testing for geographical, social or psychic
* Unilateral cervical radiotherapy Indication

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2015-12-03 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
cumulative dose of administered cisplatin in each arm | 36 months after the end of treatment
  cisplatin dose amount received at each cycle

SECONDARY OUTCOMES:
Frequency of toxicities | Every week during treatment and every 3 months after treatment up to 3 years
  Assessment of toxicity in accordance with NCI-CTC-AE 4.03
Maximum Platine Concentration [Cmax], | Cycle 1 before infusion, 90 min, 180 min,210 min, 270 min, 360 min and 420 min after the beginning of infusion in comparator arm and before infusion, 30 min, 45 min,75 min, 135 min, 225 min in experimental arm at Day 1 and Day 4
  Blood sample
Area Under the Curve [AUC] of platine | Cycle 1 before infusion, 90 min, 180 min, 210 min, 270 min, 360 min and 420 min after the beginning of infusion in comparator arm and before infusion, 30 min, 45 min, 75 min, 135 min, 225 min in experimental arm at Day 1 and Day 4
  Blood sample
Values of Neutrophil Gélatinase-associated Lipocalin (NGAL) | Baseline and 24hour after infusion of cisplatin in comparator arm and 24hour after the last infusion of cisplatin in experimental arm
  Urinary sample
Doses of radiation | 7 weeks after the beginning of radiotherapy
  total dose received
Duration of radiation | 7 weeks after the beginning of radiotherapy
  Interruption of radiotherapy due to toxicity
Loco-regional failure rate | 36 months after the end of randomization
  Delay between the date of randomisation and the occurrence of a recurrence
overall survival | 36 months after the end of randomization
  Delay between the date of randomization and death

CONTACTS AND LOCATIONS:
Overall Officials: Christian BOREL, MD, Principal Investigator — Centre Paul Strauss
Locations (1):
- Centre Paul Strauss, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Yes